CLINICAL TRIAL: NCT03526900
Title: Phase II Non-randomized Study of a Atezolizumab (MPDL3280A) in Combination With Carboplatin Plus Pemetrexed in Patients Who Are Chemotherapy-naïve and Have Stage IV Non-squamous Non-small Cell Lung Cancer Twith Asymptomatic Brain Metastasis
Brief Title: Atezolizumab in Combination With Carboplatin Plus Pemetrexed in Chemotherapy-naïve Patients With Asymptomatic Brain Metastasis
Acronym: ATEZO-BRAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 17/05_ATEZO-BRAIN; 2017-005154-11 (EudraCT Number)
Record Dates: First submitted 2018-04-18; First posted 2018-05-16 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Induction phase: atezolizumab will be given intravenously (iv) at a dose of 1200 mg for 60 minutes on day 1 of each cycle. Subsequent atezolizumab cycles may be administered for 30 minutes, if there were no perfusion-related toxicity. Pemetrexed will be administered at a dose of 500 mg/m2 IV for 15 minutes on day 1 of each cycle. In addition, folic acid, vitamin B12, and dexamethasone 4 mg will be given the day before and the day after treatment with pemetrexed. Carboplatin will be given at a dose with an area under the 5 curve for 30 minutes on day 1 of each cycle, approximately 30 minutes after the pemetrexed infusion is complete. After completing 4 to 6 cycles of Carboplatino plus pemetrexed and atezolizumab, patients will continue with pemetrexed in combination with atezolizumab (maintenance phase) until they have an unacceptable toxicity, progression of the disease, decision of the patient/physician or have Completed 2 years of treatment.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — * Induction (four or six 21-day cycles) : Atezolizumab 1200 mg / iv + carboplatin 5 AUCs + pemetrexed 500 mg/m2
  * Maintenance (21-day cycles): atezolizumab 1200 mg/iv + pemetrexed 500 mg/m2.
  Other Names: Tecentriq

SUMMARY:
This is a multicenter, national, nonrandomized, phase II trial in subjects with nonsquamous NSCLC patients that have untreated asymptomatic BM. A pre-screening period using brain MRI for patients diagnosed with advanced non-squamous NSCLC EGFR/ALK wild type and ECOG PS 0-1 will be crucial to identify patients with asyntomatic BM. Forty patients will be recruited.

DETAILED DESCRIPTION:
Atezolizumab will be administered intravenously (iv) at a dose of 1200 mg over 60 minutes on day 1 of each cycle. The subsequent cycles of atezolizumab can be administered over 30 minutes, if there were no infusion-related toxicities. Pemetrexed will be administered at a dose of 500 mg/m2 iv over 15 minutes on day 1 of each cycle. In addition, folic acid, vitamin B12, and dexamethasone 4mg bid will be administered one day before and after pemetrexed treatment. Carboplatin will be administered at a dose with an area under the curve of 5 over 30 minutes on day 1 of each cycle approximately 30 minutes after the end of the pemetrexed infusion. After completing 4 to 6 cycles of carboplatin plus pemetrexed and atezolizumab, patients will continue with pemetrexed in combination with atezolizumab until unacceptable toxicity, disease progression, patient/physician decision or completion of 2 years of therapy.

Tumor measurements by CT scan (systemic response) and brain MRI (intracranial response) will be performed every 6 weeks until the 12th week and thereafter every 9 weeks until disease progression. In case of brain progression, rescue with brain radiotherapy should be considered. In case of exclusive brain progression, patients are allowed to receive brain radiotherapy (WBRT or SRS) and then continue with study therapy if the patients maintain clinical benefit and appropriate performance status (ECOG PS≤2).Immunotherapy should be started no later than 4 weeks after completing radiation therapy (brain radiotherapy 2 weeks + 4 weeks of recovery from potential acute toxicity). In case of systemic progression without brain progression, a novel line of systemic treatment should be considered. Patients experiencing systemic progression and/or brain progression will be followed and two post-progression visits will be performed at 30 and 90 days.

Response will be assessed independently in the brain and systemically: systemic response will be evaluated according to RECIST v1.1 and brain response according to the RANO response assessment criteria for BM (RANO-BM). Adverse events will be assessed throughout and assessed using the CTCAE version 4.03. EORTC quality of life questionnaire EORTC C30 and the submodules QLQ-LC13 and BN20 will be assessed in the ITT population at baseline, cycle 5 (week 12),cycle 9 (week 24), at end of study treatment (30 and 90 days) and/or at disease progression. Periodic evaluations of the trial data will be conducted by an independent DMC to ensure subject safety and to evaluate the efficacy at the interim analyses. Neurocognitive assessment including the standardized neuropsychological tests: Hopkins Verbal Learning Test (HVLT), Trail Making Test (TMT), Rey-Osterrieth complex figure test (ROCF) and Controlled Oral Word Association Test (COWA) will be assessed at baseline cycle 5 (week 12),cycle 9 (week 24), at end of study treatment (30 and 90 days) and/or at disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Signed written informed consent.
* ECOG Performance Status (PS) of 0 to 1.
* Subjects with histologically or cytologically confirmed stage IV non-squamous NSCLC who did not received any prior chemotherapy or brain radiotherapy. Patients with EGFR mutation or ALK fusion will be excluded.
* Patients who received prior neo-adjuvant, adjuvant chemotherapy or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months since the last dose of chemotherapy and/or radiotherapy.
* Asymptomatic or oligosymptomatic(considered to have alterations in the neurological examination, whether or not they are noted in the anamnesis, that do not prevent appropriate functioning according to the patients' basal state, or that disappear with medical treatment (corticosteroids, analgesics, anticonvulsants) untreated brain metastases.
* Steroids treatment (dexamethasone) is allowed and patients that remained oligosymptomatic or asymptomatic for 2 weeks on steroids will be eligible when they were receiving ≤ 4mg dexamethasone once a day.
* Systemic measurable disease by computed tomography (CT) per response evaluation criteria in solid tumors version (RECIST) 1.1 criteria AND brain measurable disease by magnetic resonance imaging (MRI) per RANO-BM criteria.
* Availability of a formalin-fixed paraffin-embedded block (cell blocks will be accepted if tumor biopsy is not available) containing tumor tissue or 10 unstained slides.
* Adequate hematopoietic, hepatic and renal function:

ANC ≥ 1,500 cells/μL o Lymphocyte count ≥ 500 cells/μL o Platelet count ≥ 100,000 cells μL o Hemoglobin ≥ 9.0 g/dL (transfusion are is allowed) o INR or aPTT ≤ 1.5 x upper limit of normal (ULN); patients receiving therapeutic anticoagulation should be on a stable dose o ALT, AST and/or alkaline phosphatase ≤ 2.5 x ULN, with the following exceptions: -patients with known liver metastasis: ALT and/or AST ≤ 5 x ULN -patients with known bone metastasis: alkaline phosphatase ≤ 5 x ULN o Serum bilirubin ≤ 1.5 x ULN; patients with known Gilbert disease who have serum bilirubin ≤ 3 x ULN may be recruited) o Calculated creatinine clearance (CRCL) ≥ 45 mL/min (based on the standard Cockcroft and Gault formula).

* For women of childbearing potential: agreement to remain abstinent or use contraceptive non-hormonal methods with a failure rate of 1% per year during the treatment period and for 3 months after the last dose of study treatment. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of non-hormonal contraceptive methods with a failure rate of 1% per year include bilateral tubal ligation, male sterilization and copper intrauterine devices.
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm. With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 3 months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period.

Exclusion Criteria:

* History of other malignancy within 3 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* Patients harboring an EGFR mutation or an ALK fusion will be excluded
* Leptomeningeal carcinomatosis or metastases in the brain stem, mid-brain, pons, medulla or lesions causing obstructive hydrocephalus
* Patients with neurological symptoms, including those receiving > 4mg of dexamethasone will not be eligible for this study
* Spinal or hemorrhagic metastases will be excluded
* Prior surgical resection of brain or spinal lesions in the prior 14 days
* Previous systemic treatment or neo-adjuvant or adjuvant chemotherapy less than 6 months before enrollment
* Clinical significant comorbidities that impaired administration of platinum-based chemotherapy
* History of autoimmune disease, including but not limited to myasthenia gravis, myosistis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone are eligible for this study
  * Patients with controlled Type 1 diabetes mellitus on a stable dose of insulin are eligible for this study
  * Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g. patients with psoriasic arthritis would be excluded) are permitted provided that they meet the following conditions: rash covers less than 10% of body surface area, disease is well controlled at baseline and only requires lowpotency topical steroids, no acute exacerbations during the last 12 months
* History of idiopathic pulmonary fibrosis, drug-induced pneumonitis or active radiation pneumonitis out of the radiation field
* Previous treatment with immune checkpoint inhibitors or CD137 and OX-40 agonists
* Treatment with investigational therapy within 28 days prior to initiation of study drug - Positive for hepatitis C virus (HCV) antibody or for hepatitis B surface antigen (HBsAg) at screening. Patients with past or resolved hepatitis B virus (HBV) infection (HBcAb positive with absence of HBsAg) would be eligible whether they are negative for HBV DNA. Patients positive for HCV antibody would be eligible whether they are negative for HCV RNA
* Active tuberculosis or HIV infection
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Nadal, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (15):
- Spain (15):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari Germans Tries i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario de la Coruña, A Coruña, Coruña
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital General de Alicante, Alicante
  - H.U.Vall D´Hebrón, Barcelona
  - Hospital de Santa Creu i Sant Pau, Barcelona
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Fundación Jiménez Díaz, Madrid
  - H. La Paz, Madrid
  - Hospital General Universitario de Valencia, Valencia
  - Hospital La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nadal E, Rodriguez-Abreu D, Simo M, Massuti B, Juan O, Huidobro G, Lopez R, De Castro J, Estival A, Mosquera J, Sullivan I, Felip E, Blasco A, Guirado M, Pereira E, Vilarino N, Navarro V, Bruna J. Phase II Trial of Atezolizumab Combined With Carboplatin and Pemetrexed for Patients With Advanced Nonsquamous Non-Small-Cell Lung Cancer With Untreated Brain Metastases (Atezo-Brain, GECP17/05). J Clin Oncol. 2023 Oct 1;41(28):4478-4485. doi: 10.1200/JCO.22.02561. Epub 2023 Aug 21. PMID 37603816
- See also: Grupo Español de Cáncer de Pulmón website — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening details:Patients who are chemotherapy naïve and have Stage IV non-squamous NSCLC with untreated brain metastases will be enrolled in this study.
  Study enrollment was completed between November 2018 and December 2019.
Groups:
- Atezolizumab: Induction phase: atezolizumab will be given intravenously (iv) at a dose of 1200 mg for 60 minutes on day 1 of each cycle. Subsequent atezolizumab cycles may be administered for 30 minutes, if there were no perfusion-related toxicity. Pemetrexed will be administered at a dose of 500 mg/m2 IV for 15 minutes on day 1 of each cycle. In addition, folic acid, vitamin B12, and dexamethasone 4 mg will be given the day before and the day after treatment with pemetrexed. Carboplatin will be given at a dose with an area under the 5 curve for 30 minutes on day 1 of each cycle, approximately 30 minutes after the pemetrexed infusion is complete. After completing 4 to 6 cycles of Carboplatino plus pemetrexed and atezolizumab, patients will continue with pemetrexed in combination with atezolizumab (maintenance phase) until they have an unacceptable toxicity, progression of the disease, decision of the patient/physician or have Completed 2 years of treatment.
  Atezolizumab: - Induction (four or six 21-day cycles) : Atezolizumab 1200 mg / iv + carboplatin 5 AUCs + pemetrexed 500 mg/m2
  -Maintenance (21-day cycles): atezolizumab 1200 mg/iv + pemetrexed 500 mg/m2.
Period: Overall Study
Arm/Group | Atezolizumab
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population (ITT): Intention to treat analysis will include all patients that will be registered into the clinical trial.
Arm/Group | Atezolizumab
Number analyzed (Participants) | 40
Age, Continuous [Median (Standard Deviation); unit: years] | 66.75 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 40
Performance Status [Number; unit: participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  participants
    ECOG 0 | 14
    ECOG 1 | 26
    ECOG 2 | 0
    ECOG 3 | 0
    ECOG 4 | 0
Cigarrette Smoking History [Count of Participants; unit: Participants]
  Never Smoke | 6
  Former Smoke | 11
  Smoker | 23
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 39
  Adenosquamous | 0
  Squamous | 0
  Large Cell Carcinoma | 0
  NOS/Undifferentiated | 1
PD-L1 expression [Count of Participants; unit: Participants] — PD-L1 tumor proportion score expression was conducted at each center by immunohistochemical analysis after clinical practice using the Dako 22C3 and Ventana SP263 antibodies. PD-L1 expression was considered positive when ≥1% of tumor cells had PD-L1 membranous staining.
  Participants
    ≥ 50% | 10
    1%-49 % | 10
    0 % | 18
    Unknown | 2
Baseline corticosteroids [Count of Participants; unit: Participants]
  Yes | 22
  No | 18
Diagnosis of brain metastases [Count of Participants; unit: Participants]
  Synchronous | 37
  Metachronous | 3
Total number of brain lesions per patient [Median (Full Range); unit: Number of lesions] | 5 [1 to 20]
Total number of target brain lesions per patient [Median (Full Range); unit: Number of lesions] | 1 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Atezolizumab + CBDCA + Pemetrexed by Evaluating PFS Rate
Description: Percentage of subjects without disease progression (intracranial or systemic) at 12 weeks after enrollment. Determined by the investigator according to RANO and RECIST v1.1 criteria for brain and systemic disease respectively. Response Evaluation Criteria In Solid Tumors (RECIST v1.1) for target lesions and assessed by MRI:Complete Response(CR),Disappearance of all target lesions; Partial Response (PR) ≥30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD) ≥20% increase in the sum of diameters of target lesions. Reponse Evaluation criteria in brain metastasis (RANO) for target lesions assessed by MRI: Complete Response (CR) Disappearance of all CNS target lesions without use of corticosteroids, Partial response (PR) ≥30% decrease in the sum longest diameter of CNS target lesions;Progessive disease (PD) ≥20% increase in the sum longest diameter of CNS target lesions
Time Frame: 12 weeks after enrollment
Population: Intention-to-treat population cohort of 40 patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 40
percentage of participants | 62.2 [47.1 to 76.2]

2. Secondary Outcome: Efficacy of Atezolizumab + CBDCA + Pemetrexed by Measuring Objective Response.
Description: Objective response defined as a complete response or partial response on two consecutive evaluations 6 weeks apart, as determined by the investigator according to RANO and RECIST v1.1 criteria for brain and systemic disease respectively. Response Evaluation Criteria In Solid Tumors (RECIST v1.1) for target lesions and assessed by MRI: Complete Response(CR), Disappearance of all target lesions; Partial Response (PR) ≥30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD) ≥20% increase in the sum of diameters of target lesions. Reponse Evaluation criteria in brain metastasis (RANO) for target lesions assessed by MRI: Complete Response (CR), Disappearance of all CNS target lesions without use of corticosteroids, Partial response (PR) ≥30% decrease in the sum longest diameter of CNS target lesions; Progessive disease (PD) ≥20% increase in the sum longest diameter of CNS target lesions or the appearance of new lesions
Time Frame: Two consecutive evaluations 6 weeks apart
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 40
Participants | 18

3. Other Pre Specified Outcome: Overall Response by RANO Criteria and Steroids
Description: To record the number of patients best response with steroid vs without steroid. Response Evaluation criteria in brain metastasis (RANO-BM) for target lesions and assessed by MRI: Complete Response (CR) Disappearance of all CNS target lesions, Partial response (PR) ≥30% decrease in the sum longest diameter of CNS target lesions; Overall Response (OR) = CR + PR. Progessive disease (PD) ≥20% increase in the sum longest diameter of CNS target lesions or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months.
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 38
Participants
  No steroids Stable disease or progression | 11
  No steroids Complete response or partial response | 7
  Yes steroids Stable disease or progression | 10
  Yes steroids Complete response or partial | 10

4. Other Pre Specified Outcome: Median Time to Brain Radiotherapy (WBRT or SRS)
Description: Register the median time to needed brain radiotherapy (WBRT or SRS).
Time Frame: From date of randomization until the date of first needed salvage therapy, assessed up to 48 months.
Population: Per protocol population
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 24
months | 10.9 [7.8 to 15.9]

ADVERSE EVENTS:
Time Frame: 48 months
Description: The severity of AE will be determined using CTCAE version 4.03
Arm/Group | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 28/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=40)
Nephritis (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Pulmonary embolism (Vascular disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=40)
Anemia (General disorders) | 8 (8)
Fatigue (General disorders) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Anorexia (General disorders) | 4 (4)
Platelet count decreased (Blood and lymphatic system disorders) | 3 (3)
Alanine aminotransferase increased (Hepatobiliary disorders) | 2 (2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lipase increased (Hepatobiliary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03526900/Prot_SAP_000.pdf